CLINICAL TRIAL: NCT01409915
Title: Pilot Phase 2 Trial of the Safety & Efficacy of Granulocyte-Macrophage Colony-Stimulating Factor (Leukine®) in the Treatment of Alzheimer's Disease
Brief Title: Study of the Safety & Efficacy of Leukine® in the Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Dana Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-1273
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; neuropsychological assessment; Granulocyte-Macrophage Colony-Stimulating Factor; Leukine
MeSH Terms: conditions — Alzheimer Disease | interventions — Colony-Stimulating Factors; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sagramostim (Leukine) (Experimental): 5 subjects 250 mcg /m2/day Leukine subcutaneously for 5 days/week for three weeks. Data and Safety Monitoring Board will then review data and recommend whether to continue at the same current recommended dose for additional subjects or to reduce the dose by half if excessive leukocytosis occurs
  Interventions: Drug: Sagramostim
- Control Group (Placebo Comparator): Saline -- placebo comparator. Given as a subcutaneous injection.
  Interventions: Drug: Saline -- placebo comparator

INTERVENTIONS:
Drug: Sagramostim — 5 subjects 250 mcg /m2/day Leukine subcutaneously for 5 days/week for three weeks. Data and Safety Monitoring Board will then review data and recommend whether to continue at the same current recommended dose for additional subjects or to reduce the dose by half if excessive leukocytosis occurs
  Other Names: Leukine; Granulocyte-Macrophage Colony-Stimulating Factor
  Arms: Sagramostim (Leukine)
Drug: Saline -- placebo comparator — subcutaneous injection
  Other Names: Sterile solution of sodium chloride in water
  Arms: Control Group

SUMMARY:
A medicine that is FDA-approved for bone marrow stimulation (called Leukine) will be tested for its ability to be tolerated by Alzheimer's disease patients and potentially to improve their memory.

DETAILED DESCRIPTION:
Preliminary preclinical results demonstrated that GM-CSF (Granulocyte macrophage colony-stimulating factor, e.g. Leukine®/Sargramostim) rapidly reduced cerebral amyloid deposition and completely reversed memory deficits in transgenic mouse models of Alzheimer's Disease (AD). To assess the efficacy of GM-CSF in humans, the investigators performed a retrospective analysis of a cognition study of human patients undergoing hematopoietic cell transplantation for cancer and who garner cognitive impairments from the chemotherapy or irradiation. In the patients that received a colony-stimulating factor (CSF) to stimulate the bone marrow and recover immune system function, the investigators found that those who received GM-CSF (Leukine®/Sargramostim) plus G-CSF (Filigrastim) significantly improved in cognitive function as compared to those who received G-CSF alone. These findings combined with over two decades of accrued safety data using recombinant human GM-CSF, Leukine®/Sargramostim, in elderly leukopenic patients, suggested that Leukine® should be tested as a treatment to reverse cerebral amyloid pathology and cognitive impairment in AD.

ELIGIBILITY:
Inclusion Criteria:

1. age 55 to 85 years;
2. should have a mild-to-moderate AD diagnosis (MMSE 10-26 inclusive);
3. should have evidence of elevated cortical amyloid by PET using florbetapir F18 (Amyvid) [i.e. a positive scan], assessed qualitatively according to the Amyvid product label.
4. if on anti-dementia treatment should be on stable treatment for at least 2 months (i.e. cholinesterase inhibitor and/or Memantine or Axona);
5. stable on all other medications for at least 30 days prior to screen;
6. should be fluent in English;
7. should be physically able to participate by medical history, clinical exam and tests;
8. should have a study partner to accompany them to scheduled visits.

Exclusion Criteria:

1. clinically relevant arrhythmias;
2. a resting pulse less than 50;
3. active cancer other than non-melanoma skin cancers;
4. use of another investigatory drug within 2 months of screening;
5. significant stroke or head trauma by history or MRI;
6. contraindication for having a MRI;
7. diagnostic and Statistical Manual of Mental Disorders-IV criteria for a current major psychiatric disorder;
8. sensitivity to yeast or yeast products;
9. impaired kidney function as measured by a Glomerular Filtration Rate less than 60 milliliters/min;
10. preexisting fluid retention, pulmonary infiltrates, or congestive heart failure;
11. history of moderate-to-severe lung disease;
12. history of moderate-to-severe liver disease;
13. pregnant women, or any women who feel they are likely to become pregnant during the study;
14. prisoners.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huntington Potter, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sagramostim (Leukine): 250 mcg /m2/day Leukine subcutaneously for 5 days/week for three weeks.
- Control Group: Saline placebo comparator: subcutaneous injection
Period: Overall Study
Arm/Group | Sagramostim (Leukine) | Control Group
Started | 21 | 23
Completed | 20 | 20
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is Per Protocol, with all participants enrolled and randomized in the clinical trial, and who complete the treatment without major breaches in the study protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sagramostim (Leukine) | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.10 (6.57) | 70.15 (6.42) | 68.63 (6.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: White / Caucasian | 20 | 19 | 39
  Race / Ethnicity: Black / African American | 0 | 1 | 1
  Race / Ethnicity: Asian / Pacific Islander | 0 | 0 | 0
  Race / Ethnicity: Hispanic / Latino | 0 | 0 | 0
  Race / Ethnicity: Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Education Level (Mean years) [Mean (Standard Deviation); unit: Years] | 15.70 (2.92) | 15.80 (2.71) | 15.75 (2.78)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) by Body System
Description: Count of AE's from Consent to Follow-up 2 within a safety analysis set consisting of all participants who were enrolled and randomized and who received at least one injection of sargramostim or placebo
Time Frame: 20 weeks (From Consent to Follow-up 2)
Population: Safety analysis set (SAS), all participants enrolled and randomized and who received at least one injection of sargramostim or placebo
Measure: Number; unit: Adverse Events
Arm/Group | Sagramostim (Leukine) | Control Group
Number analyzed (Participants) | 21 | 22
Adverse Events
  Cardiovascular AE | 5 | 2
  Constitutional | 6 | 5
  Dental | 1 | 0
  Dermatological | 16 | 5
  ENT | 2 | 0
  Gastrointestinal | 8 | 5
  Musculoskeletal | 8 | 11
  Neurological | 9 | 2
  Psychological | 0 | 2
  Respiratory | 4 | 4

2. Secondary Outcome: MMSE (Mini Mental State Examination) From Baseline to End of Treatment (3 Weeks), Follow-Up 1 (45 Days Post Treatment) and Follow-Up 2 (90 Days Post Treatment)
Description: Mini-Mental State Examination (MMSE) is a brief psychometric instrument developed to assess cognitive function in elderly populations. It is a standard assessment used by all NIH Alzheimer's Disease Centers (ADCCs and ADRCs) to identify and monitor individuals with AD. The range for scores in the MMSE is from 0 to 30, with lower scores indicating greater impairment.
Time Frame: From Baseline to End of Treatment (3 weeks), Follow-Up 1 (45 days post treatment) and Follow-Up 2 (90 days post treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sagramostim (Leukine) | Control Group
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 17.10 (4.57) | 20.75 (4.97)
  End of Treatment (3 weeks) | 18.55 (4.99) | 20.40 (5.28)
  Follow-up 1 (45 days post treatment) | 18.00 (5.52) | 19.90 (5.19)
  Follow-up 2 (90 days pot treatment) | 17.10 (5.78) | 19.40 (5.47)

3. Secondary Outcome: Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) From Baseline to End of Treatment (3 Weeks), Follow-Up 1 (45 Days Post Treatment) and Follow-Up 2 (90 Days Post Treatment)
Description: Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-Cog13). The ADAS-Cog13 is the most popular cognitive testing instrument used in clinical trials of nootropics (drugs or agents that improve cognitive function). It consists of 13 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities, which are often referred to as the core symptoms of AD. Score ranges from 0-85, with a higher score representing more severe impairment
Time Frame: Baseline to End of Treatment (3 weeks), Follow-Up 1 (45 days post treatment) and Follow-Up 2 (90 days post treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sagramostim (Leukine) | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 43.20 (12.45) | 36.20 (12.01)
  End of Treatment (3 weeks) | 43.54 (12.02) | 36.68 (11.63)
  Follow-up 1 (45 days post treatment) | 47.67 (11.89) | 36.33 (9.85)
  Follow-up 2 (90 days post treatment) | 45.87 (13.21) | 36.85 (10.24)

4. Other Pre Specified Outcome: Alzheimer's Disease Cooperative Study -Activities of Daily Living Inventory (ADCS-ADL) From Baseline to End of Treatment (3 Weeks), Follow-Up 1 (45 Days Post Treatment) and Follow-Up 2 (90 Days Post Treatment)
Description: The ADCS-ADL is a caregiver/study partner rated questionnaire of 23 items, with possible scores over a range of 0-78, where 78 implies full functioning with no impairment. The ADCS-ADL assesses functional capacity across a wide spectrum of severity
Time Frame: Baseline to End of Treatment (3 weeks), Follow-Up 1 (45 days post treatment) and Follow-Up 2 (90 days post treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sagramostim (Leukine) | Control Group
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 56.50 (12.30) | 62.75 (8.98)
  End of Treatment (3 weeks) | 57.00 (11.93) | 61.85 (9.32)
  Follow-up 1 (45 days post treatment) | 53.35 (14.02) | 59.85 (9.05)
  Follow-up 2 (90 days post treatment) | 53.30 (15.00) | 60.30 (9.00)

5. Other Pre Specified Outcome: Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) From Baseline to End of Treatment (3 Weeks), Follow-Up 1 (45 Days Post Treatment) and Follow-Up 2 (90 Days Post Treatment)
Description: The CDR is a study partner/caregiver and participant based interview to assess changes in domains such as memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated as 0 (no dementia), 0.5 (uncertain dementia), 1 (mild dementia), 2 (moderate dementia), or 3 (severe dementia). The Sum of Boxes score (CDR-SB) score was tallied for each administration using the rules from the Washington University Knight ADRD scoring algorithm. Scores range from 0-18. The higher the score, the worse the impairment.
Time Frame: Baseline to End of Treatment (3 weeks), Follow-Up 1 (45 days post treatment) and Follow-Up 2 (90 days post treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sagramostim (Leukine) | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 7.10 (3.32) | 6.10 (2.67)
  End of Treatment (3 weeks) | 7.53 (3.37) | 5.95 (2.37)
  Follow-up 1 (45 days post treatment) | 8.42 (4.22) | 6.81 (3.12)
  Follow-up 2 (90 days post treatment) | 8.57 (4.14) | 7.03 (3.27)

6. Other Pre Specified Outcome: Trail Making Test - Part A (TMT-A) From Baseline to End of Treatment (3 Weeks), Follow-Up 1 (45 Days Post Treatment) and Follow-Up 2 (90 Days Post Treatment)
Description: The Trail Making Test- part A (TMT-A) is a assessment of psychomotor speed and is a timed test in which participants must connect a series of numbers randomly placed on a page. Time range is between 0 and 150 seconds, with higher score representing worse performance.
Time Frame: Baseline to End of Treatment (3 weeks), Follow-Up 1 (45 days post treatment) and Follow-Up 2 (90 days post treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sagramostim (Leukine) | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 101.50 (46.17) | 84.85 (48.83)
  End of Treatment (3 weeks) | 92.60 (45.49) | 79.40 (44.56)
  Follow-up 1 (45 days post treatment) | 107.85 (45.81) | 84.00 (45.64)
  Follow-up 2 (90 days post treatment) | 110.35 (45.55) | 85.45 (48.10)

ADVERSE EVENTS:
Time Frame: Adverse events were completed over a 20 week period, from Consent to Follow-up 2
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Sagramostim (Leukine) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/23
Other Adverse Events (participants affected / at risk) | 19/21 | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sagramostim (Leukine) (N=21) | Control Group (N=23)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sagramostim (Leukine) (N=21) | Control Group (N=23)
Fatigue (General disorders) | 2 | 4
Injection site reaction (Skin and subcutaneous tissue disorders) | 9 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 3
Pain/Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Fall (Musculoskeletal and connective tissue disorders) | 1 | 4
Headache, Benign NOS (Nervous system disorders) | 8 | 2
Upper Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
The main weakness is the small sample size of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT01409915/Prot_SAP_000.pdf